CLINICAL TRIAL: NCT04575194
Title: Cardiovascular and Metabolic Effects of Drugs for the Treatment of Obesity
Brief Title: Study of the Cardiometabolic Effects of Obesity Pharmacotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Athens Medical Center (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obesity drugs study
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Blood Pressure
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Naltrexone-Bupropion combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide 3 mg (Active Comparator): Patients will be prescribed sc liraglutide 3 mg/day along with a dietary and physical activity intervention.
  Interventions: Drug: Liraglutide 6 MG/ML [Saxenda]
- Naltrexone/bupropion 32/360 mg (Active Comparator): Patients will be prescribed oral naltrexone/bupropion 32/360 mg/day along with a dietary and physical activity intervention.
  Interventions: Drug: Naltrexone-Bupropion Combination

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML [Saxenda] — 3 mg of sc liraglutide daily plus lifestyle intervention
  Arms: Liraglutide 3 mg
Drug: Naltrexone-Bupropion Combination — 32/360 mg of oral lnaltrexone-bupropion daily plus lifestyle intervention
  Arms: Naltrexone/bupropion 32/360 mg

SUMMARY:
The aim of the present study is to compare the efficacy of liraglutide vs. naltrexone/bupropion on metabolic and cardiovascular risk markers, weight loss, as well as the postprandial secretion of gastrointestinal hormones involved in hunger and satiety, after a test meal. The study will include 40 patients, who will further be divided into two treatment groups (20 patients on liraglutide vs. 20 patients on naltrexone/bupropion). The patients will be examined at baseline, 3 and 6 months after the treatment initiation.

DETAILED DESCRIPTION:
This is a prospective study of patients aged ≥18 years, who are overweight (BMI ≥ 27 kg / m2 in the presence of dyslipidemia or hypertension or obstructive sleep apnea or fatty infiltration or prediabetes) or obese patients (BMI ≥ 30 kg / m2). Patients' data will be collected before starting medication (time 0) and at 3 and 6 months under treatment in the clinical practice of the selected drug, as described in the drug's package leaflet, along with a simultaneous dietary intervention and exercise. Patient groups will be comparable in age, gender and BMI.

The aim of the study is the comparison of the efficacy of liraglutide vs. naltrexone/bupropion in metabolic and cardiovascular markers.

The following parameters will be measured:

* Weight, height, waist and hip circumference
* 24-hour recording of blood pressure and heart rate
* HbA1c, total cholesterol, LDL, HDL, urine albumin/creatinine ratio
* Bioelectric impedance for determination of total and visceral fat and muscle mass Indirect calorimetry for the determination of resting metabolic rate and total energy expenditure
* Determination of baroreflex sensitivity (BRS) and heart rate variability (HRV) to investigate the function of the autonomic nervous system
* Blood sample test meal at 0, 30, 60, 90, 120, 150 and 180 min to determine insulin concentration and gastrointestinal hormones involved in hunger and satiety with modern indirect calorimetry to determine postprandial thermogenic analog scales (VAS)
* Neuropathy tests
* Assessment of quality of life with the SF-36 questionnaire and assessment of the feeling of hunger and satiety
* Echocardiographic determination of the left systolic and telodiastolic diameter of the left ventricle, cardiac fat and the Tei index at times 0 and 6 months with medication
* Pericardial fat

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with BMI ≥ 30 kg / m2 or BMI ≥ 27 kg / m2 in the presence of dyslipidemia or hypertension or obstructive sleep apnea or fatty infiltration or prediabetes.

Exclusion Criteria:

1. Presence of any clinical contraindications for the administration of liraglutide or bupropion / naltrexone
2. Bariatric surgery
3. Diabetes type 2
4. Active malignancy
5. Medication that affects weight (eg corticosteroids, phenothiazines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure | 3 and 6 months
  Blood pressure as assessed by 24-hour recording (numerical scale)

SECONDARY OUTCOMES:
Weight loss | 3 and 6 months
  Percentage of weight lost will be measured by an electronic scale (numerical scale)
Changes in glycemic | 3 and 6 months
  Measurement of HbA1c will be measured biochemically (numerical scale)
Changes in lipemic profile | 3 and 6 months
  Total cholesterol, Triglycerides, LDL-C, HDL-C will be measured biochemically (numerical scale)
Percentage of visceral fat | 3 and 6 months
  Measurement of visceral fat by bioimpedance analysis (numerical scale)
Fat mass | 3 and 6 months
  Measurement of fat mass by bioimpedance analysis (numerical scale)
Fat free mass | 3 and 6 months
  Measurement of fat free mass by bioimpedance analysis (numerical scale)
Autonomic nervous system function | 3 and 6 months
  Measurement of heart rate variability will be measured through Ewing score and Spectral analysis testing (numerical scale)
Changes in meal induced thermogenesis | 3 and 6 months
  Measurement through indirect calorimetry and assessment of changes in Resting Metabolic Rate (RMR) (numerical scale)
Changes in gut hormones involved in appetite regulation | 3 and 6 months
  Measurement in plasma before and after the intervention during a mixed meal test will be measured through ELISA kits (numerical scale)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- First Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stefanakis K, Kokkinos A, Simati S, Argyrakopoulou G, Konstantinidou SK, Kouvari M, Kumar A, Kalra B, Mantzoros CS. Circulating levels of all proglucagon-derived peptides are differentially regulated postprandially by obesity status and in response to high-fat meals vs. high-carbohydrate meals. Clin Nutr. 2023 Aug;42(8):1369-1378. doi: 10.1016/j.clnu.2023.06.026. Epub 2023 Jun 28. PMID 37418844